CLINICAL TRIAL: NCT04524104
Title: Study of a PST-Trained Voice-Enabled Artificial Intelligence Counselor (SPEAC) for Adults With Emotional Distress (Phase 1)
Acronym: SPEAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Penn State University (Other); Washington University School of Medicine (Other); Stanford University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Beth and George Vitoux Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-0918; 1R61MH119237-01A1 (NIH)
Record Dates: First submitted 2020-08-14; First posted 2020-08-24 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumen treatment (Experimental): Participants will complete functional magnetic resonance imaging (fMRI) and self-report questionnaires at baseline and 16 weeks. Participant will receive an encrypted study iPad enabled with Lumen at baseline. They will complete 8 PST sessions beginning with 4 weekly and then 4 biweekly intervals (i.e., on weeks 1, 2, 3, 4, 6, 8, 10, 12) over 12 weeks on their assigned iPad. Participants will also complete naturalistic end-of-day assessments for 7 days every 2 weeks (on weeks 0, 2, 4, 6, 8, 10, 12, 16), that is, 8 time series. Additionally, participants will complete depressive and anxiety symptoms questionnaire and user experience surveys at all PST sessions.
  Interventions: Behavioral: Lumen Treatment
- Waitlist Control (No Intervention): Participants will complete functional magnetic resonance imaging (fMRI) and self-report questionnaires at Baseline and 16 weeks.
  Participant will receive an encrypted study iPad at baseline. Participants will complete naturalistic end-of-day assessments for 7 days every 2 weeks (on weeks 0, 2, 4, 6, 8, 10, 12, 16), that is, 8 time series.
  Participants in the waitlist control arm will only complete assessments but will have the option to receive Lumen at the end of the study. The PST module on the study iPad will be disabled until their 16-week assessment is completed, at which time they will have the option to complete 8 PST sessions on their assigned iPads.

INTERVENTIONS:
Behavioral: Lumen Treatment — the virtual AI agent, Lumen, via an iPad-based application. Each participant will receive a locked, encrypted study iPad installed with Lumen. They will complete 8 problem solving therapy (PST) sessions beginning with 4 weekly and then 4 biweekly intervals over 12 weeks on their assigned iPad.
  Arms: Lumen treatment

SUMMARY:
In the phase 1 of the SPEAC project the specific aims are to: (1) establish the functionality, usability, and treatment fidelity of Lumen using iterative, user-centered design, development, and formative evaluation; and (2) demonstrate feasibility, acceptability, and target engagement in a 2-arm pilot RCT. The aim 1 focuses on developing a voice-enabled, artificial intelligence (AI) virtual agent, named Lumen, trained in Problem Solving Therapy (PST) via an iPad-based application. The development of Lumen will employ iterative user-centered design-evaluation cycles. After the functionality, usability and treatment fidelity of Lumen are established, in the aim 2, we will conduct a 2-arm randomized clinical trial (RCT, Study 1) to pilot test Lumen.

DETAILED DESCRIPTION:
60 participants with eligible depression and/or anxiety (n=60) will be randomized in a 2:1 ratio to the Lumen treatment arm (n=40) or the wait-list control arm (n=20).

Participants in both arms will receive encrypted study iPads.

Lumen treatment arm participants will receive encrypted study iPads to complete PST with Lumen (8 sessions, 4 weekly and then 4 biweekly, over 12 weeks) or be on a wait list. Participant permission will be obtained to record their PST sessions with Lumen, which will be independently rated by PST experts for fidelity. Lumen treatment arm participants will also complete the depressive and anxiety symptoms assessment questionnaires at the start of each PST session, and a participant survey of usability, user experience and therapeutic alliance at the end of each PST session.

Participants in both arms will complete measurements of neural target engagement and treatment outcomes at both baseline (0 week) and 16 weeks.

These assessments will include (1) functional magnetic resonance imaging (fMRI) 2) Surveys of PST (3) Surveys of patient-reported outcomes, such as depressive and anxiety symptoms, social functioning, and health-related quality of life. Participants also will complete naturalistic end-of-day assessments of mood, stress, appraisal, and coping for 7 days every 2 weeks (on weeks 0, 2, 4, 6, 8, 10, 12, 16) - that is, 8 time series.

Participants in the wait-list control arm will have the option to receive Lumen at the end of the study. The PST module on the study iPad will be disabled until their 16-week assessment is completed, at which time they will have the option to complete 8 PST sessions on their assigned iPads.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at study enrollment
* Emotional distress defined by elevated depressive (PHQ9 scores 10-19) and/or anxious symptoms (GAD7 scores 10-14)
* Willing and able to provide written informed consent and HIPAA authorization

Exclusion Criteria:

* Unable to speak, read, understand English for informed consent (grade 6 level)
* Current pharmacotherapy or psychotherapy (individual or professionally-led group therapy) for depression or anxiety
* Suicidal ideation per PHQ9 with active plan
* Bipolar or psychotic disorder, or current psychiatric treatment
* Weight ≥350 pounds due to brain scanner constraints, MRI contraindications, traumatic brain injuries, and tumor or any other known structural abnormality in the brain
* Severe medical condition (e.g., myocardial infarction or stroke or new cancer diagnosis in the past 6 months, end-stage organ failure, terminal illness) or residence in a long-term care facility
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past year
* Active alcohol or substance use disorder (including prescription drugs) based on the CAGE Questionnaire Adapted to Include Drugs (CAGE-AID)
* Cognitive impairment based on the Callahan 6-item screener
* Current or planned pregnancy or lactating (<6 months postpartum)
* Participation in other investigational treatment studies that would significantly affect participation in this study, raise safety concerns, and/or confound outcomes (participant may be asked to provide the informed consent of the other study for final decision on exclusion by a study psychiatrist)
* Family/household member of an already enrolled participant or of a study team member
* Plan to move out of the Chicagoland area during the study period
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Department of Medicine, Vitoux Program on Aging and Prevention, Chicago, Illinois
  - UIMC Advanced Imaging Center, Chicago, Illinois

REFERENCES:
- [Derived] Lv N, Kannampallil T, Xiao L, Ronneberg CR, Kumar V, Wittels NE, Ajilore OA, Smyth JM, Ma J. Association Between User Interaction and Treatment Response of a Voice-Based Coach for Treating Depression and Anxiety: Secondary Analysis of a Pilot Randomized Controlled Trial. JMIR Hum Factors. 2023 Nov 6;10:e49715. doi: 10.2196/49715. PMID 37930781

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumen Treatment | Waitlist Control
Started | 42 | 21
Completed | 40 | 21
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumen Treatment | Waitlist Control | Total
Number analyzed (Participants) | 42 | 21 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.9) | 35.6 (11.5) | 37.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 15 | 43
  Male | 14 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 15 | 7 | 22
  African American | 8 | 8 | 16
  Asian/Pacific Islander | 5 | 2 | 7
  Hispanic | 12 | 3 | 15
  Other (e.g., declined to state, multirace) | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 42 | 21 | 63
HADS Depression score [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS), including 7 questions for anxiety and 7 questions for depression, measures self-reported anxiety and depression in a general medical population of patients. Each item on the questionnaire is scored from 0-3 and the score for either anxiety or depression ranges between 0 and 21 with the following categories: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Total score for the entire scale (emotional distress) ranges from 0 to 42, with higher score indicating more distress.
  units on a scale | 7.6 (2.9) | 6.7 (3.2) | 7.3 (3.0)
HADS Anxiety score [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS), including 7 questions for anxiety and 7 questions for depression, measures self-reported anxiety and depression in a general medical population of patients. Each item on the questionnaire is scored from 0-3 and the score for either anxiety or depression ranges between 0 and 21 with the following categories: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Total score for the entire scale (emotional distress) ranges from 0 to 42, with higher score indicating more distress.
  units on a scale | 11.0 (2.7) | 9.9 (4.1) | 10.6 (3.3)
HADS Total score [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS), including 7 questions for anxiety and 7 questions for depression, measures self-reported anxiety and depression in a general medical population of patients. Each item on the questionnaire is scored from 0-3 and the score for either anxiety or depression ranges between 0 and 21 with the following categories: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Total score for the entire scale (emotional distress) ranges from 0 to 42, with higher score indicating more distress.
  units on a scale | 18.6 (4.3) | 16.6 (6.6) | 17.9 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Activation of Left Amygdala From Baseline Functional Magnetic Resonance Scan at 16 Weeks
Description: Two neural targets defined a priori, specifically activation of the amygdala for nonconscious threat-related emotional reactivity and activation of the DLPFC for cognitive control will be assessed using fMRI. In the facial emotion viewing paradigm, facial expression stimuli are standardized black and white photographs of 8 identities (4 female, 4 male) with evoked expressions of threat-related emotions (fear, anger), sad-related emotions (sadness) and reward-related emotions (happiness), along with neutral. To assess amygdala activation for the negative affect circuit, our analysis focused on threatening faces only. Threat stimuli included a combination of fear and anger stimuli relative to neutral blocks. For the Go-NoGo paradigm, the 'Go' and 'NoGo' stimuli are presented for 500 ms each with an inter-stimulus interval of 750 ms. Higher score indicates higher activation of the amygdala and DLPFC.
Time Frame: Baseline, 16 weeks
Population: The number of participants in the Participant Flow module reflects number of participants who provided any data (e.g., HADS data) at 16 weeks. Among them, 30 Lumen Intervention participants and 19 Waitlist Control participants had quality fMRI data at 16 weeks.
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 30 | 19
beta weights | -0.07 (0.39) | -0.13 (0.29)

2. Primary Outcome: Change in Activation of Right Amygdala From Baseline Functional Magnetic Resonance Scan at 16 Weeks
Description: as for outcome 1
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 30 | 19
beta weights | -0.14 (0.44) | -0.07 (0.40)

3. Primary Outcome: Change in Activation of Left dlPFC From Baseline Functional Magnetic Resonance Scan at 16 Weeks
Description: as for outcome 1
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 30 | 19
beta weights | -0.02 (0.49) | 0.09 (0.43)

4. Primary Outcome: Change in Activation of Right dlPFC From Baseline Functional Magnetic Resonance Scan at 16 Weeks
Description: as for outcome 1
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 30 | 19
beta weights | -0.10 (0.64) | 0.09 (0.78)

5. Secondary Outcome: Change From Baseline Hospital Anxiety and Depression Scale (HADS) Depression Score at 16 Weeks
Description: HADS, including 7 questions for anxiety and 7 questions for depression, measures self-reported anxiety and depression in a general medical population of patients. Each item on the questionnaire is scored from 0-3 and the score for either anxiety or depression ranges between 0 and 21 with the following categories: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Total score for the entire scale (emotional distress) ranges from 0 to 42, with higher score indicating more distress. Cronbach's alpha coefficients range from 0.78-0.93 for the anxiety subscale and from 0.82-0.90 for the depression subscale. Test-retest correlations are ≥0.80 after ≤2 weeks. Correlations of the anxiety and depression subscales with commonly used anxiety and depression measures (e.g., Beck Depression Inventory, Patient Health Questionnaire, State-Trait Anxiety Inventory, Symptom Checklist-90-Revised) vary between 0.60 (good) and 0.80 (very good).
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -1.85 (4.00) | 0.10 (3.95)

6. Secondary Outcome: Change From Baseline Hospital Anxiety and Depression Scale (HADS) Anxiety Score at 16 Weeks
Description: as for outcome 5
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -2.25 (4.48) | 0.14 (5.11)

7. Secondary Outcome: Change From Baseline Hospital Anxiety and Depression Scale (HADS) Total Score at 16 Weeks
Description: as for outcome 5
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -4.10 (7.53) | 0.24 (8.49)

8. Secondary Outcome: Change From Baseline Social Problem-Solving Inventory-Revised: Short Form (SPSI-R:S) at 16 Weeks
Description: Participants' problem solving abilities will be assessed using the reliable and valid SPSI-R:S that contains 25 items in the following 5 subscales: positive problem orientation (PPO), negative problem orientation (NPO), rational problem solving (RPS), impulsive/careless style (ICS), and avoidance style (AS). Each item is rated on a 5-point scale ranging from "not at all true of me" (0) to "extremely true of me" (4). The SPSI-R:S assessed total problem-solving ability. The total problem-solving ability score ranged from 0 to 20 by averaging the subscale scores, with the higher score indicating more productive problem-solving skills.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | 0.83 (2.92) | 0.42 (2.19)

9. Secondary Outcome: Change From Baseline Dysfunctional Attitudes Scale (DAS) at 16 Weeks
Description: DAS (Form A) is a 40-item self-reported scale that measures the presence and intensity of dysfunctional attitudes. Each item is rated a 7-point Likert scale (7 = fully agree; 1 = fully disagree). DAS score is the sum of the 40 items, with a range of 40-280. Higher score indicates the more dysfunctional attitudes an individual possesses.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -12.8 (30.39) | -6.62 (20.49)

10. Secondary Outcome: Change From Baseline Penn State Worry Questionnaire (PSWQ) at 16 Weeks
Description: PSWQ is a self-reported, 16-item, Likert-type scale that measures the trait of worry. PSWQ score has a range of 16-80, with a higher total score indicating more worry.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -3.90 (9.99) | -3.95 (11.01)

11. Secondary Outcome: Change From Baseline Positive Affect Score of the Positive and Negative Affect Schedule (PANAS) at 16 Weeks
Description: PANAS consists of two 10-item self-reported scales to measure positive and negative affect. Each item asks about the extent one has felt a positive or negative feeling on a 5-point scale of 1 (not at all) to 5 (very much). Positive Affect scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | 4.03 (7.79) | 2.43 (7.89)

12. Secondary Outcome: Change From Baseline Negative Affect Score of the Positive and Negative Affect Schedule (PANAS) at 16 Weeks
Description: PANAS consists of two 10-item self-reported scales to measure positive and negative affect. Each item asks about the extent one has felt a positive or negative feeling on a 5-point scale of 1 (not at all) to 5 (very much). Negative Affect scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -1.60 (9.67) | -0.90 (7.58)

13. Secondary Outcome: Change From Baseline Sheehan Disability Scale at 16 Weeks
Description: The Sheehan Disability Scale is a validated questionnaire that measures functional disability and is sensitive to treatment effects in clinical trials. Cronbach's alpha is 0.89. Patients rate the extent to which their symptoms impair work/school, social, and family life on a visual analog scale from 0 (Not at all) to 10 (Extremely) and answer the number of days when their symptoms cause them to miss work/school and be unproductive at work/school. Total score is the sum of the three separate scores on work/school, social, and family life, ranging from 0 to 30.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | -3.70 (10.50) | -2.00 (6.94)

14. Secondary Outcome: Change From Baseline Percent Work Time Missed Due to Health at 16 Weeks
Description: Work productivity and activity impairment questionnaire (WPAI) consists of 6 questions and measures impairments in work and activities. Four main outcomes can be calculated and expressed in percentages by multiplying the scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for people who were currently employed; 2) percent impairment while working due to health = Q5/10 for people who were currently employed and actually worked in the past 7 days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for people who were currently employed; and 4) percent activity impairment due to health Q6/10 for all respondents.
Time Frame: Baseline, 16 weeks
Population: Some participants among the responders at baseline and 4 months were not currently employed. The overall number of participants analyzed was less than 40 Lumen participants and 21 Control participants.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 32 | 16
percentage of work time missed | 5.08 (22.22) | 0.29 (16.12)

15. Secondary Outcome: Change From Baseline Percent Impairment While Working Due to Health at 16 Weeks
Description: as for outcome 14
Time Frame: Baseline, 16 weeks
Population: Among the responders (40 Lumen participants and 21 Control participants), only those who were currently employed and actually worked in the past 7 days were included in analysis.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 28 | 15
percentage of impairment while working | -13.21 (33.12) | -7.33 (28.65)

16. Secondary Outcome: Change From Baseline Percent Overall Work Impairment Due to Health at 16 Weeks
Description: as for outcome 14
Time Frame: Baseline, 16 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 32 | 16
percentage of overall work impairment | -8.82 (36.13) | -8.76 (32.56)

17. Secondary Outcome: Change From Baseline Percent Activity Impairment Due to Health at 16 Weeks
Description: as for outcome 14
Time Frame: Baseline, 16 weeks
Population: At baseline 41 out of 62 participants did not provide response to this question.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 15 | 7
percentage of activity impairment | 9.33 (32.83) | 2.86 (16.04)

18. Secondary Outcome: Change From Baseline Physical Health Composite Score of the 12-item Short-Form Health Survey (SF12) at 16 Weeks
Description: The SF-12 is a 12-item version of the SF-36 that measures overall health-related quality of life. Physical and mental health composite scores are computed using the scores of 12 questions and range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health. Test-retest correlation is 0.89 for the physical health subscale and 0.76 for the mental health subscale.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | 1.37 (6.95) | -0.21 (7.30)

19. Secondary Outcome: Change From Baseline Mental Health Composite Score of the 12-item Short-Form Health Survey (SF12) at 16 Weeks
Description: as for outcome 18
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 40 | 21
score on a scale | 3.57 (9.93) | 2.09 (9.47)

20. Secondary Outcome: Change From Baseline Daily Mood (Positive Affect) at 16 Weeks
Description: Daily end-of-day assessments will be captured over a one-week period at baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 16). During active treatment in the Lumen arm (Studies 1 & 2) or the in-person PST arm (Study 2), this will occur for 3 days prior to, the day of, and for 3 days after a scheduled PST session. For waitlist controls, this will occur for 7 days starting on Sunday of each assigned week. Daily mood will be measured using 8 mood items (0 = Not at all, 6 = Extremely), with 4 measuring positive affect and 4 measuring negative affect. Positive affect score is mean of item scores, with higher scores indicating more positive affect. Negative affect score is mean of item scores, with higher scores indicating more negative affect.
Time Frame: From Baseline to every 2 week, up to 16 weeks
Population: Among Lumen and Control participants, 34 and 18 had provided data at both baseline and 16 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 34 | 18
score on a scale | 0.27 (0.97) | -0.50 (0.91)

21. Secondary Outcome: Change From Baseline Daily Mood (Negative Affect) at 16 Weeks
Description: as for outcome 20
Time Frame: From Baseline to every 2 week, up to 16 weeks
Population: Among Lumen and Control participants, 34 and 18 had provided data at both baseline and 16 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 34 | 18
score on a scale | -0.55 (0.72) | -0.07 (1.10)

22. Secondary Outcome: Change From Baseline Daily Stress at 16 Weeks
Description: Daily end-of-day assessments will be captured over a one-week period at baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 16). During active treatment in the Lumen arm (Studies 1 & 2) or the in-person PST arm (Study 2), this will occur for 3 days prior to, the day of, and for 3 days after a scheduled PST session. For waitlist controls, this will occur for 7 days starting on Sunday of each assigned week. Daily stress will be assessed by the question "how stressful was your day today" (0 = Not at all, 6 = Extremely).
Time Frame: From Baseline to every 2 weeks, up to 16 weeks
Population: Among Lumen and Control participants, 34 and 18 had provided data at both baseline and 16 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 34 | 18
score on a scale | -0.95 (1.03) | -0.15 (1.12)

23. Secondary Outcome: Change From Baseline Daily Appraisal at 16 Weeks
Description: Daily end-of-day assessments will be captured over a one-week period at baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 16). During active treatment in the Lumen arm (Studies 1 & 2) or the in-person PST arm (Study 2), this will occur for 3 days prior to, the day of, and for 3 days after a scheduled PST session. For waitlist controls, this will occur for 7 days starting on Sunday of each assigned week. The appraisal items will focus on assessing "problem orientation" or the general awareness and appraisals of problems during the day. A main appraisal question asks "To what degree were you able to accept your problem as normal or an expected part of everyday life?" (0 = Not at all, 6 = A great deal).
Time Frame: From Baseline to every 2 weeks, up to 16 weeks
Population: Among Lumen and Control participants, 34 and 18 had provided data at both baseline and 16 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 34 | 18
score on a scale | 0.05 (1.34) | -0.26 (0.89)

24. Secondary Outcome: Change in Depression Symptoms From First PST Session in Week 1 to Eighth Session in 12 Weeks
Description: PHQ-9 is a self-administered instrument for screening, diagnosing, monitoring, and measuring the severity of depression. It rates the frequency of symptoms as "0" (not at all) to "3" (nearly every day) and has been validated for use in primary care. The PHQ-9 total score ranges from 0 to 27 and is categorized as follows: None or minimal depression 0-4, Mild depression 5-9, Moderate depression 10-14, Moderately severe depression 15-19, and Severe depression 20-27. Cronbach's alpha coefficients range from 0.86 to 0.89 and test-retest correlations range from 0.84-0.95 within 48 hours and from 0.81-0.96 at 7-day reassessment. PHQ-9 scores were found to be highly correlated with Beck Depression Inventory scores in the general population (r=0.73).
Time Frame: From start of first PST session in week 1 to week (2, 3, 4, 6, 8, 10, 12) up to 12 weeks
Population: Among 40 Lumen participants and 21 Control participants, 34 and 16 completed PHQ-9 at both session 1 and session 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 34 | 16
score on a scale | -3.41 (4.85) | -0.25 (4.39)

25. Secondary Outcome: Change in Anxiety Symptoms From First PST Session in Week 1 to Eighth Session in 12 Weeks
Description: GAD-7 is a valid and reliable 7-question scale to screen for 4 anxiety disorders: Post Traumatic Stress Disorder, Panic Disorder, Generalized Anxiety Disorder, and Social Phobia. A score of ≥10 indicates a high probability of 1 or more of these disorders. Cronbach's alpha is 0.92 and test-retest correlation is 0.83. GAD-7 scores also correlate highly with scores of 2 commonly-used anxiety scales: the Beck Anxiety Inventory (r=0.72) and the anxiety subscale of the Symptom Checklist-90 (r=0.74).
Time Frame: From start of first PST session in week 1 to week (2, 3, 4, 6, 8, 10, 12) up to 12 weeks
Population: Among 40 Lumen participants and 21 Control participants, 34 and 18 completed GAD-7 at both session 1 and session 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 34 | 18
score on a scale | -3.15 (4.70) | -1.61 (5.90)

26. Secondary Outcome: Change in NASA Task Load Index (TLX) From First PST Session in Week 1 to Eighth Session in 12 Weeks
Description: A modified version of the NASA Task Load Index (TLX) measures workload. The TLX rating sheet was administered assuming similar weights for each of the 5 task load items: mental demand, temporal demand (e.g., being rushed), effort, frustration, and performance. The original TLX includes a physical demand item which was not included herein, as it was not applicable for the task of interacting with Lumen. An overall task load index score was calculated as sum of the 5 task load items, each ranging from 1 to 7. A higher overall score reflected greater (unfavorable) demand.
Time Frame: From end of first PST session in week 1 to week (in week, 2, 3, 4, 6, 8, 10, 12) up to 12 weeks
Population: Only Lumen participants completed NASA Task Load Index (TLX) and 24 Lumen participants completed TLX at both session 1 and session 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 24 | 0
score on a scale | 2.21 (8.28) |

27. Secondary Outcome: Change in User Experience Questionnaire-Short Version (UEQ-S) From First PST Session in Week 1 to Eighth Session in 12 Weeks
Description: UEQ-S is a validated instrument containing 8 items from the 26 items of the original UEQ. UEQ-S measures user experience. From the UEQ-S survey, scale values were calculated by rescaling the survey responses to the range -3 to 3 and UEQ-S total score were calculated as mean of survey responses. UEQ-S total scores <-0.8 represented a negative evaluation, between -0.8 and 0.8 represented a neutral evaluation, and >0.8 represent a positive evaluation.
Time Frame: From end first PST session in week 1 to week (in week 2, 3, 4, 6, 8, 10, 12) up to 12 weeks
Population: Only Lumen participants completed Experience Questionnaire-Short version (UEQ-S) and 24 Lumen participants completed UEQ-S at both session 1 and session 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 24 | 0
score on a scale | -0.17 (1.10) |

28. Secondary Outcome: Change in Adapted Working Alliance Inventory for Digital Coaching Interventions (WAI-Tech) From First PST Session in Week 1 to Eighth Session in 12 Weeks
Description: WAI-Tech was based closely on the original 36-item WAI and uses a parallel set of 36 items rated on a 7-point scale (1 = "never" to 7 = "always") to measure the level of alliance between patient and digital coach along 3 domains: Task (12 items), Bond (12 items), and Goal (12 items). An overall score was calculated based on item means. A higher overall score reflected a greater treatment alliance.
Time Frame: From end of first PST session in week 1 to week (in week 2, 3, 4, 6, 8, 10, 12) up to 12 weeks
Population: Only Lumen participants completed Adapted Working Alliance Inventory for digital coaching interventions (WAI-Tech) and 24 Lumen participants completed WAI-Tech at both session 1 and session 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumen Treatment | Waitlist Control
Number analyzed (Participants) | 24 | 0
score on a scale | -0.15 (0.94) |

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Lumen Treatment | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/42 | 2/21
Other Adverse Events (participants affected / at risk) | 9/42 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumen Treatment (N=42) | Waitlist Control (N=21)
Gastrointestinal system (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reproductive system (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Neurological system (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumen Treatment (N=42) | Waitlist Control (N=21)
Hematological system (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Musculoskeletal system (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Reproductive system (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Neurological (Nervous system disorders) | 1 (1) | 1 (1)
Gastrointestinal system (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal/Urologic system (Renal and urinary disorders) | 0 (0) | 1 (1)
Immunologic system (Immune system disorders) | 0 (0) | 1 (1)
General disorders (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04524104/Prot_SAP_000.pdf